CLINICAL TRIAL: NCT06909019
Title: The Menu Labels for Environmental Impact and Nutrition Study (MENU Study): Online Experiment
Brief Title: MENU Study: Online Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of California, Davis (Other); Harvard School of Public Health (HSPH) (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00027451; 1R01DK139327-01 (NIH)
Record Dates: First submitted 2025-03-26; First posted 2025-04-03 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Food Selection
Keywords: food labeling; climate labeling; choice behavior
MeSH Terms: conditions — Food Preferences | interventions — Product Labeling

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to view two fast-food menus presented in random order with one of five labeling schemes applied: (1) a QR code on all items (control); (2) a low climate impact label on all low impact items (3) a high climate impact label on high impact items; (4) traffic light labels on all items by level of impact; and (5) climate grade labels on all items by level of impact. All fast-food menus will include main items, sides, desserts, and drinks. Labels will only appear alongside main menu items and will be assigned using thresholds for greenhouse gas emissions set a priori in kilograms of CO2 equivalent per kilogram of food. Participants will be instructed to select a hypothetical lunch meal order. The investigators will record participant meal selections and, using publicly available nutritional information for each item selected, calculate a score of overall meal healthfulness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (QR) Labels (Placebo Comparator): A black label featuring a QR code and white text that reads "SCAN HERE" will be placed beneath all main menu items on two restaurant menus. Explanatory text describing the label's meaning will be displayed at the top of the menu.
  Interventions: Behavioral: Control (QR) Labels
- Low Climate Impact Labels (Experimental): A green icon-plus-text label that reads "LOW CLIMATE IMPACT" in white text against a green background will be placed on two restaurant menus beneath main menu items with a low climate impact using a predetermined threshold of estimated greenhouse gas emissions set at <2.6 kgCO2e. Labels will include a white globe icon directly preceding the label text. Explanatory text describing the label's meaning will be displayed at the top of the menu.
  Interventions: Behavioral: Low Climate Impact Labels
- High Climate Impact Labels (Experimental): A red icon-plus-text label that reads "HIGH CLIMATE IMPACT" in white text against a red background will be placed on two restaurant menus beneath main menu items with a high climate impact using a predetermined threshold of estimated greenhouse gas emissions set at >=9.2 kgCO2e. Labels will include a white globe icon directly preceding the label text. Explanatory text describing the label's meaning will be displayed at the top of the menu.
  Interventions: Behavioral: High Climate Impact Labels
- Traffic Light Labels (Experimental): Traffic Light labels will be placed on two restaurant menus beneath all main menu items. Using predetermined estimated greenhouse gas emission thresholds, each item will be assigned one of three icon-plus-text labels within this scheme: low-, medium-, or high-impact label, set in kgCO2e at <2.6, >=2.6 & <9.2, and >=9.2, respectively. Each will read, "HIGH CLIMATE IMPACT" within a red label, "MED. CLIMATE IMPACT" in a yellow label, and "LOW CLIMATE IMPACT" in a green label. Text for all labels written in white, and a white globe icon will precede the text. Explanatory text describing the meaning of the labels will be displayed at the top of the menu.
  Interventions: Behavioral: Traffic Light Labels
- Climate Grade Labels (Experimental): Climate Grade labels will be placed on two restaurant menus beneath all main menu items, using predetermined estimated greenhouse gas emission thresholds to assign one of five icon-plus-text labels which indicate a specific climate impact grade (A, B, C, D, and F). Thresholds are set in kgCO2e as follows: [A] <1.7, [B] >=1.7 & <2.6, [C] >=2.6 & <9.2, [D] >=9.2 & <28, [F] >=28. All labels are solid black with a white globe icon followed by white text which reads "CLIMATE GRADE". On the left side of each label, a grade is displayed, capitalized and in a white font within a solid-colored box. The color of the box corresponds with each letter grade: A = dark green, B = light green, C = yellow, D = orange, F = red. Beneath the letter grade, a gradient of all possible grades is displayed horizontally in smaller font, each grade atop a small solid box in the respective grade color. Explanatory text describing the meaning of the labels will be displayed at the top of the menu.
  Interventions: Behavioral: Climate Grade Labels

INTERVENTIONS:
Behavioral: Control (QR) Labels — Participants will view two fast-food restaurant menus presented in a random order. Each menu will include main, side, dessert, and drink items, and each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, Control (QR) labels will be displayed beneath each item. Participants will be instructed to select at least 1 and up to 4 menu items for a hypothetical meal order. Participants will be required to select a main item and, optionally, up to 3 additional items (drinks, sides, desserts).
  Arms: Control (QR) Labels
Behavioral: Low Climate Impact Labels — Participants will view two fast-food restaurant menus presented in a random order. Each menu will include main, side, dessert, and drink items, and each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, Low Climate Impact labels will be displayed beneath each item. Participants will be instructed to select at least 1 and up to 4 menu items for a hypothetical meal order. Participants will be required to select a main item and, optionally, up to 3 additional items (drinks, sides, desserts).
  Arms: Low Climate Impact Labels
Behavioral: High Climate Impact Labels — Participants will view two fast-food restaurant menus presented in a random order. Each menu will include main, side, dessert, and drink items, and each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, High Climate Impact labels will be displayed beneath select items. Participants will be instructed to select at least 1 and up to 4 menu items for a hypothetical meal order. Participants will be required to select a main item and, optionally, up to 3 additional items (drinks, sides, desserts).
  Arms: High Climate Impact Labels
Behavioral: Traffic Light Labels — Participants will view two fast-food restaurant menus presented in a random order. Each menu will include main, side, dessert, and drink items, and each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, Traffic Light labels will be displayed beneath each item. Participants will be instructed to select at least 1 and up to 4 menu items for a hypothetical meal order. Participants will be required to select a main item and, optionally, up to 3 additional items (drinks, sides, desserts).
  Arms: Traffic Light Labels
Behavioral: Climate Grade Labels — Participants will view two fast-food restaurant menus presented in a random order. Each menu will include main, side, dessert, and drink items, and each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, Climate Grade labels will be displayed beneath each item. Participants will be instructed to select at least 1 and up to 4 menu items for a hypothetical meal order. Participants will be required to select a main item and, optionally, up to 3 additional items (drinks, sides, desserts).
  Arms: Climate Grade Labels

SUMMARY:
The primary objective of this study is to test the relative effects of climate-impact menu label designs on the healthfulness of consumers' fast-food meal choices. Participants will complete hypothetical online meal ordering tasks using a survey which emulates the online menus of two types of fast-food chain restaurants: a burger restaurant and a sandwich restaurant. Participants will be randomized the view both menus, presented in random order, with one of five labeling conditions applied. Secondary objectives include examining total greenhouse gas emissions per meal order, energy and nutrient content of meals ordered, prices of meals ordered, and, through a post-order survey, noticeability, and perceptions, and knowledge and understanding of labels between the conditions.

DETAILED DESCRIPTION:
This online randomized trial will test the relative effects of climate impact menu label designs on the healthfulness of consumers' fast-food meal choices and perceptions of menu items. The survey research firm National Opinion Research Center (NORC) will recruit a nationally representative sample of 6,000 adults aged 18 years and older who speak English and reside in the United States from the Center's AmeriSpeak Panel.

Participants will complete a between-subjects online experiment in which the participants will be randomized to view two fast-food online ordering menus (in randomized order) with one of five labeling schemes applied: (1) a QR code on all items (control); (2) a low climate impact label on all low impact items (3) a high climate impact label on high impact items; (4) traffic light labels on all items by level of impact; and (5) climate grade labels on all items by level of impact. Each restaurant menu will be presented across 2 pages; page 1 will display all main items, and page 2 will display categories for side, dessert, and drink items. Labels will only appear alongside main menu items and will be assigned using thresholds for greenhouse gas emissions set a priori in kilograms of carbon dioxide (CO2) equivalent per kilogram of food. Each hypothetical order must include between 1 and 4 items. Participants will be required to select 1 main item and, optionally, up to 3 additional items (drinks, sides, desserts). After completing the meal ordering task, participants will be prompted to answer questions about the whether the participant noticed the correct label for the participant's condition, whether the participant used the label when making meal selections, perceptions of the labeled menu items and the labeling condition which the participants were randomized to view, knowledge of the relative climate impact of food items and consumer behaviors, and support of governmental and policies and practices regarding food and nutrition. Additionally, participants will be asked about level of food security, use of GLP-1 agonists, personal values, dietary patterns, and other demographic information. Participation in the study will last approximately 10 minutes.

The primary outcome will be the healthfulness of meal orders selected from the online menu, indicated by a modified Nutrient Profile Index meal score for all food items ordered. Secondary outcomes will be total greenhouse gas emissions per meal ordered, total calories ordered, whether a sugar-sweetened beverage was ordered, and perceived message effectiveness of the climate-impact labels.

Analyses will be conducted overall (summing the meal selections across both restaurants) and stratified by restaurant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Member of the NORC AmeriSpeak Panel
* Residing in the United States

Exclusion Criteria:

* <18 years of age
* Not residing in the United States
* Completed the survey in less than one-third of the median completion duration of all participants
* Respondents with high refusal rates (skipped or refused more than 50% of questions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6294 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Modified Nutrient Profile Index score | During online survey ordering task, up to 10 minutes
  Healthfulness of fast-food meal selections, measured with a modified Nutrient Profile Index (NPI) score. NPI scores are based on the United Kingdom (UK) Ofcom Nutrient Profiling Model, which is used to score individual foods in the UK to determine which ones can be marketed to children. The NPI is a 0 to 100-point score for foods; a score of >=64 is considered healthy. NPI awards points from nutrients to encourage (e.g., fiber, protein) and nutrients of concern (e.g., sodium, sugar) per 100 grams. The investigators will generate a modified NPI score to evaluate the healthfulness of full meals comprised of multiple food items. This measure will be determined by calculating the weighted mean NPI score of all food items selected per meal, with each item's NPI score weighted by its proportionate contribution of mass in grams to the total mass of the meal. Beverages are excluded and assessed through secondary outcomes.

SECONDARY OUTCOMES:
Nutrient Profile Index score | During online survey ordering task, up to 10 minutes
  The healthfulness of the fast-food main item selections, measured with a Nutrient Profile Index (NPI) score. NPI scores are based on the United Kingdom (UK) Ofcom Nutrient Profiling Model, which is used to score individual foods in the UK to determine which ones can be marketed to children. The NPI is a 0 to 100-point score for foods; a score of >=64 is considered healthy. NPI awards points from nutrients to encourage (e.g., fiber, protein) and nutrients of concern (e.g., sodium, sugar) per 100 grams.
Total greenhouse gas emissions | During online survey ordering task, up to 10 minutes
  Cumulative total kilograms of carbon equivalent (kgCO2e) per kilogram of food for all meal items. Beverages are excluded and assessed through other secondary outcomes. Beverages are excluded and assessed through secondary outcomes (#5 & #11).
Frequency of red meat selected | During online survey ordering task, up to 10 minutes
  Measured as a dichotomous variable (yes/no) indicating whether participants' hypothetical meal orders include an item containing red meat.
Total energy selected (number of calories) | During online survey ordering task, up to 10 minutes
  The total number of calories in participants' hypothetical meal orders, calculated as the sum of calories across all menu items selected. Higher values indicate more calories selected.
Total amount of saturated fat (grams) selected | During online survey ordering task, up to 10 minutes
  The total amount of saturated fat in participants' hypothetical meal orders, calculated as the sum of saturated fat (grams) across all menu items selected. Higher values indicate more saturated fat selected.
Total amount of sugar (grams) selected | During online survey ordering task, up to 10 minutes
  The total amount of sugar in participants' hypothetical meal orders, calculated as the sum of sugar (grams) across all menu items selected. Higher values indicate more sugar selected.
Total amount of protein (grams) selected | During online survey ordering task, up to 10 minutes
  The total amount of protein in participants' hypothetical meal orders, calculated as the sum of protein (grams) across all menu items selected. Higher values indicate more protein selected.
Total amount of fiber (grams) selected | During online survey ordering task, up to 10 minutes
  The total amount of fiber in participants' hypothetical meal orders, calculated as the sum of fiber (grams) across all menu items selected. Higher values indicate more fiber selected.
Total amount of sodium (milligrams) selected | During online survey ordering task, up to 10 minutes
  The total amount of sodium in participants' hypothetical meal orders, calculated as the sum of sodium (milligrams) across all menu items selected. Higher values indicate more sodium selected.
Frequency of sugar-sweetened beverage selected | During online survey ordering task, up to 10 minutes
  Measured as a dichotomous variable (yes/no) indicating whether participants' hypothetical meal orders include a sugar-sweetened beverage.
Percentage of participants with knowledge of the climate impact of foods | During online survey post-ordering task, up to 10 minutes
  This outcome will measure participants' knowledge of the relative climate impacts of meals with different main proteins. Participants are prompted to numerically rank three meals by climate impact. The exact prompt is: "Please rank the below food options from smallest (1) to largest (3) climate impact. Write "1" next to the food option with the smallest climate impact, "2" next to the option with the middle climate impact, and "3" next to the option with the largest climate impact." Each rank item reads "Meal in which the main protein is beef", "Meal in which the main protein is chicken", and "Meal in which the main protein is tofu". Responses will be analyzed by % who correctly rank the 3 items by experimental condition.
Percentage of participants with knowledge of the climate impact of menu items | During online survey post-ordering task, up to 10 minutes
  This outcome will measure participants' knowledge of the relative climate impacts of menu items by label condition. Via two questions, one per restaurant, participants are prompted to indicate "Which menu item below has a larger contribution to climate change (i.e., produces more greenhouse gas emissions)?". Three response options are provided: two images of main menu items by label condition and "The menu items have the same climate impact". Responses will be analyzed as the % who answer both questions correctly by label condition.
Frequency of participants with attention to labels | During online survey post-ordering task, up to 10 minutes
  Measured by whether participants noticed labels on the menus, in addition to calorie labels. The exact question is, "On the menus you saw, did you notice any labels (other than calories) next to or below the menu items?" Response options are "Yes", "No", and "Don't Know".
Frequency of participants who recall labels that also correctly identify purpose of labels | During online survey post-ordering task, up to 10 minutes
  Measured by whether participants who noticed labels, in addition to calorie labels, correctly identify the purpose of the labels. Response options are "Sugar", "Sodium", "QR code", "Climate Impact", "Organic", "Healthy", "Unhealthy", "None of these", and "I don't know/ I can't remember".
Perceived message effectiveness (PME) as assessed by the University of North Carolina (UNC) PME scale | During online survey post-ordering task, up to 10 minutes
  This modified 4-item UNC-PME scale measures how much the label placed beneath high climate impact menu items, discouraged consumption or evoked concern or unpleasantness about consumption of high climate impact foods. Responses to all questions will be measured on a 5-point unipolar Likert scale from 1=Not at all to 5= A great deal. The higher the score, the higher the perceived effectiveness.
Total price of meal order | During online survey ordering task, up to 10 minutes
  Measured by the cumulative total price (USD) of participants' hypothetical meal orders per restaurant, based on the prices displayed on the survey menus.
Perceived level of appeal of food items | During online survey post-ordering task, up to 10 minutes
  Measured by the level of appeal attributed to 8 main menu items, 4 from each restaurant, by label condition. All items are assessed on a 7-point Likert scale with response options of "Very unappealing", "Unappealing", "Slightly unappealing", "Neither appealing nor unappealing", "Slightly appealing", "Appealing", "Very appealing" for each food item. Higher score, higher appeal.
Perceived level of healthfulness of food items | During online survey post-ordering task, up to 10 minutes
  Measured by the level of healthfulness attributed to 8 main menu items, 4 from each restaurant, by label condition. All items are assessed on a 7-point Likert scale with response options of "Very unhealthy", "Unhealthy", "Slightly unhealthy", "Neither unhealthy nor healthy", "Slightly healthy", "Healthy," "Very healthy" for each food item.
Perceived level of climate impact of food items | During online survey post-ordering task, up to 10 minutes
  Measured by the level of climate impact attributed to 8 main menu items, 4 from each restaurant, by label condition. All items are assessed on a 7-point Likert scale with response options of "Extremely high climate impact", "Very high climate impact", "High climate impact", "Moderate climate impact", "Low climate impact", "Very low climate impact", "Extremely low climate impact" for each food item.

OTHER OUTCOMES:
Participant's knowledge of the climate impact of consumer behaviors as assessed by survey | During online survey post-ordering task, up to 10 minutes
  This outcome will measure participants' knowledge of the effectiveness of specific consumer behaviors on reducing climate change. The exact behaviors presented are: "Eat less red meat", "Eat organic foods", "Eat local, seasonal foods", "Drive less", "Use less plastic", "Save energy at home", "Recycle", "Eat fewer dairy products", "Waste less food", and "Use reusable grocery bags". Response options are: "Not effective at all", "Slightly effective", "Moderately effective", "Very effective", Extremely effective" "I don't know".
Participant's level of support for food and nutrition policies as assessed by survey | During online survey post-ordering task, up to 10 minutes
  Measured by the level of support or opposition for policies and practices regarding food, nutrition, and consumer information. This outcome is measured across five survey items with response options of "Strongly oppose", "Oppose" Somewhat oppose", "Neither support nor oppose", "Somewhat support", "Support", "Strongly support" for each specific policy described.

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Wolfson, PhD MPP, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Reimold AE, Falbe J, Kim BF, Musicus AA, Carr N, Santo R, Cho C, Leung CW, Roberto CA, Wolfson JA. The impact of restaurant menu eco labels on consumer meal selections: a randomized controlled trial. Am J Prev Med. 2026 Jan 9:108265. doi: 10.1016/j.amepre.2026.108265. Online ahead of print. PMID 41520993